CLINICAL TRIAL: NCT04871659
Title: Attitudes Behavior and Practices of Mothering Among an Online Panel
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Einhorn Family Charitable Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAAR8405
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Tantrum; Relation, Family; Parent-Child Relations; Parenting
Keywords: MTurk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online Survey completion — Eligible participants will complete surveys electronically via Amazon's mTurk platform

SUMMARY:
Subjects are users on Amazon's Mechanical Turk (MTurk) platform. MTurk users will be asked to complete a screening survey about family structure. The purpose of the screening survey is to identify MTurk users who are biological mothers of children aged 1.5 to 6 years old, and to collect survey information on how mothers interact with their children, with the aim of better understanding family relationships.

DETAILED DESCRIPTION:
This is a feasibility study that aims to identify a panel of biological mothers of children aged 1.5 to 6 years old from an online pool of participants on Amazon's Mechanical Turk (MTurk; www.mturk.com). MTurk is a novel method to recruit participants from online behavioral studies. Although MTurk workers are anonymous, demographic surveys from previous studies conducted on the web platform indicate that the majority of MTurk users are females living in the U.S. The participant pool may be of scientific interest in pursuing studies that investigate patterns of behaviors and other information pertaining to mothers. A panel of mothers that fit screening criteria may be helpful for future planned studies on attitudes, behavior, and practices surrounding mothering. The MTurk mothers panel will be eligible to participate in future studies involving knowledge, attitudes, and practices of their motherhood and of emotional connection with their children.

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers of children between ages 1.5-6 living in the US

Exclusion Criteria:

* Not having reliable internet access

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Biological mothers of children between ages 0-5 living in the US who are users of Amazon's mTurk platform
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Correlations between survey items | Day 1
  Descriptive statistics and correlations will be generated to show the basic participant characteristics captured during the data collection and whether the survey items correlate with each other. Survey items include the Parental Burnout Assessment, the Temper Loss Scale, and two surveys created by Dr. Welch at the Nurture Science Program: the Welch Emotional Connection Screen-Parent Report, as well as a tantrum questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G. Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No